CLINICAL TRIAL: NCT06466343
Title: Immunohistopathologic Findings of Cesarean Scar Niche
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelnasser Galal, Assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-05-06MD
Record Dates: First submitted 2024-06-10; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Cesarean Scar Niche
Keywords: cesarean scar, Niche

STUDY DESIGN:
Intervention Model Description: Study will be conducted on non-pregnant women with symptomatic uterine scar niche after lower segment CS at Obstetrics and Gynecology department at Sohag University Hospitals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- symptomatic non pregnant women (Other): Operative hysteroscopy will be used for surgical treatment in the cases. Hysteroscopic management of niche will be done according to the following steps: Operative procedure will be done postmenstrual, cervical preparation will be done by giving the patients misoprostol (misotac®) 400mcg two hours preoperative. Surgically, operative resectoscope (KARL STORZ, Germany,27 Fr gauge) will be inserted into the uterine cavity after cervical dilatation by Hegar uterine dilator up to 8. Distilled water will be used as distension media. Using a resectoscope, the lower edge of the niche will be trimmed, the base will be coagulated by using monopolar cutting current at 30-50 MHz.
  Interventions: Procedure: hysteroscopic resection of lower edge of cesarean scar niche

INTERVENTIONS:
Procedure: hysteroscopic resection of lower edge of cesarean scar niche — Operative hysteroscopy will be used for surgical treatment in the cases. Hysteroscopic management of niche will be done according to the following steps: Operative procedure will be done postmenstrual, cervical preparation will be done by giving the patients misoprostol (misotac®) 400mcg two hours preoperative. Surgically, operative resectoscope (KARL STORZ, Germany,27 Fr gauge) will be inserted into the uterine cavity after cervical dilatation by Hegar uterine dilator up to 8. Distilled water will be used as distension media. Using a resectoscope, the lower edge of the niche will be trimmed, the base will be coagulated by using monopolar cutting current at 30-50 MHz.
  The resected parts will be submitted together as one sampled specimen in one container of formaldehyde 30% (dissolved 800 ml water and 200 ml formaldehyde)

SUMMARY:
Niche is iatrogenic pouch like defect, present on the uterine isthmus' anterior wall where a previous caesarean section scar was made. Still, a niche has generally been defined as the myometrium's depression of at least 2 mm (Lumbanraja et al., 2024).

The literature is lacking in information about the accurate histopathologic characteristics of cesarean scar niche ridges that have been removed by hysteroscopy, as well as what critical findings to highlight and what gynaecologists can anticipate from pathology reports of cesarean scar niche specimens (AbdullGaffar & Almulla ,2022).

In this study the aim of the work is to study the histopathologic findings in cesarean scar niche specimens repaired by hysteroscopy in our institution, identify the causes of local thinning of the uterine scar after c-section to direct gynecologists regarding the efficacy of their hysteroscopic corrective repair of cesarean scar niche concerning the amelioration of symptoms, restoration of fertility, and patient follow-up.

DETAILED DESCRIPTION:
Subjects & Methods Study will be conducted on non-pregnant women with symptomatic uterine scar niche after lower segment CS at Obstetrics and Gynecology department at Sohag University Hospitals.

Patient recruitment:

All eligible patients attending at the Obstetrics and Gynecology outpatient clinic at the department will be approached by the attending physician A through explanation about the nature of the study to each patient. All patients agreeing to participate in the study will be asked to sign the informed written consent before enrollment in the study.

Ultrasound examination:

Uterine scar niche will be diagnosed by transvaginal Logic P7, GE US (frequency 50/60Hz) postmenstrual. In longitudinal plane of the uterus at anterior wall at site of CS, the depth, width, and residual myometrial thickness will be measured. All measures will be done by single operator.

Niche is iatrogenic pouch like defect, present on the uterine isthmus' anterior wall where a previous caesarean section scar was made.The myometrium's depression of at least 2 mm.

Operative procedure:

For every patient, related clinical data will be gathered, age, parity, clinical presentation, number of previous CSs, history of secondary infertility, history of previous niche repair surgeries, and follow-up data will be included in this.

Operative hysteroscopy will be used for surgical treatment in the cases.

Histopathological examination:

The hematoxylin and eosin (H&E) slides will be inspected to identify any changes related to the mucosa as well as the types of lining mucosa of the resected edges, the types of stroma and stroma-associated changes, the presence of myometrial tissue, and scarring. Slides will be also screened for inflammatory, hemorrhagic, degenerative changes, foreign body giant cell reaction and Masson trichrome stain: for staining of fibrosis (Higuchi et al., 2022).

Immunohistochemistry:

Using a sliding microtome, all paraffin-embedded blocks will be cut into 4-µm-thick sections. The parts will be floated in a water bath at 42°C before being put on slides. The antigens will be recovered in an antigen retrieval reagent following deparaffinization, CD3: a marker for T lymphocyte, CD20: a marker for B lymphocytes and CD34: a marker for angiogenesis.

Follow up:

Patients will be asked to come after 3 months for asking about improvement of symptoms, quality of life, transvaginal US evaluation will be done, and a questionnaire will be filled out (Herdman et al.,2003)

Statistical analysis:

The collected data was organized, tabulated, and statistically analyzed using Statistical Package for Social Science (SPSS) version 16 (SPSS Inc, USA). For quantitative data, mean and standard deviation (SD) will be calculated and for comparison between two means, the students (t) test will be used. For qualitative data, the frequency and percent distribution will be calculated and for comparison between groups, chi square (X2) will be used. For interpretation of results p value will be significant if less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Any Women with history of previous CS once or more with period more than one year from the last CS and had CS scar defect diagnosed by TVUS.

Exclusion Criteria:

* All women diagnosed with pelvic inflammatory disease, suspected with gynecological malignancy, postmenopausal women, women with heart disease, liver disease, renal impairment or bleeding tendency will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the incidence and type of different pathological variations within examined CS niche specimens. | three weeks
  measure the incidence and type of different pathological variations within examined CS niche specimens.

SECONDARY OUTCOMES:
correlation of predominant pathological variation with symptoms of patient and radiological findings. | 2 weeks
  estimate correlation of predominant pathological variation with symptoms of patient and radiological findings.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Ab Galal, A.lecturer, Principal Investigator — sohag faculty of medicine sohag university
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No